CLINICAL TRIAL: NCT02925130
Title: Beta2-mimetic and Central Nervous System: Effects of Salbutamol on Cortical Excitability and Cerebral Activation
Brief Title: Beta2-mimetic and Central Nervous System
Acronym: BETACTIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 38RC14339
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-03

CONDITIONS: Adrenergic Beta-2 Agonist Effect; Albuterol Effect
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Inhaled Salbutamol (Experimental): Acute inhalation of 800 microgram Salbutamol
  Interventions: Drug: Salbutamol
- Oral Salbutamol (Experimental): Acute oral intake of 4 mg Salbutamol
  Interventions: Drug: Salbutamol
- Placebo (Placebo Comparator): Acute oral intake of a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salbutamol — Acute intake of Albuterol, a beta2-mimetic, either inhaled or oral.
  Other Names: Albuterol
  Arms: Inhaled Salbutamol; Oral Salbutamol
Drug: Placebo — Acute oral intake of a placebo drug
  Other Names: Albuterol
  Arms: Placebo

SUMMARY:
Beta2-mimetics such as Salbutamol have been shown to have ergogenic effects. Acute and chronic inhaled or oral doses of Salbutamol have been shown to increase whole body exercise and muscle performances. The underlying mechanisms are however unclear. Some data suggest that Salbutamol may have some effects on the central nervous system which may explain the improved exercise and neuromuscular performances. The present study aims to assess the effects of acite inhaled or oral Salbutamol intake on the neuromuscular system by using neurostimulation techniques and magnetic resonance imaging.

DETAILED DESCRIPTION:
The effects of Salbutamol intake will be assessed by using transcranial magnetic stimulation on one hand and magnetic resonance imaging on the other hand. Maximal voluntary activation and cerebral activation will be measured during motor tasks performed until exhaustion after acute inhaled slabutamol intake, acture oral salbutamol intake or oral placebo intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without respiratory and cordiovascular diseases
* Male
* Age between 18 and 35
* Trained subjects (>6 hours of physical activity per week)
* Non- or ex-smoker (smoking cessation since at least 1 year)

Exclusion Criteria:

* Respiratory, cardiovascular and metabolic diseases
* Neuromuscular diseases
* thyrotoxicosis, or diabetes treated with insulin
* alcoholism
* MRI contraindication
* TMS contraindication

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10; Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Maximal voluntary activation | Measured immediatly after treatment intake (within 1 h)
  Measurement performed by using transcranial magnetic stimulation, superimposed on submaximal and maximal quadricep contractions

SECONDARY OUTCOMES:
Cortical activation | Measured immediatly after treatment intake (within 1 h)
  Measurement performed by using magnetic resonance imaging and the intensity of the BOLD signal in response to a motor task.
Exercise endurance | Measured immediatly after treatment intake (within 1 h)
  Time to exhaustion during the exercise muscle test.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Guinot, MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No